CLINICAL TRIAL: NCT00572819
Title: Does Self-Administered Vaginal Misoprostol Result in Cervical Ripening in Postmenopausal Women After 14 Days Pre-Treatment With Estradiol?
Brief Title: Hysteroscopy After Pretreatment With Misoprostol and Estradiol Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Britt-Ingjerd Nesheim, Gynaecological Department, Ullevål University Hospital, Oslo, Norway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-004083-52; 2007-004083-52
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Cervical Ripening
Keywords: Hysteroscopy; Misoprostol; Postmenopausal women; Cervical ripening; Dilatation; Sequential trial; Estradiol
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 1000 micrograms of self-administered vaginal misoprostol compared to placebo 12 hours before operative hysteroscopy after two weeks pretreatment with 25 micrograms daily vaginal oestradiol.
  Arms: Misoprostol
Drug: Placebo — Vaginal lactosum monohydricum administered 24 hours in postmenopausal women, compared to misoprostol after two weeks pretreatment with 25 micrograms daily vaginal oestradiol.
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether 1000 micrograms of self-administered vaginal misoprostol 12 hours before operative hysteroscopy results in effective preoperative cervical ripening after two weeks pretreatment with 25 micrograms daily vaginal estradiol, compared to placebo (lactosum monohydricum) in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* All postmenopausal (> one year since last menstruation) women who are referred to outpatient hysteroscopy with a medical indication for hysteroscopy, and who have given informed consent, will be eligible for study recruitment

Exclusion Criteria:

* Women who do not wish to participate
* Women who are medically unfit for hysteroscopy
* Women who are medically unfit for participation in any clinical trial
* Women who do not have a medical indication for hysteroscopy
* Women who have previously had, or currently have breast or gynaecological cancer
* Women who have a medical contraindication for locally applied oestradiol
* Women who are currently using hormone therapy
* Women who are unable to communicate in Norwegian, and
* Women with a known allergy to misoprostol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the preoperative baseline cervical dilatation in the two treatment groups. | 24 hours

SECONDARY OUTCOMES:
Difference between baseline cervical dilatation at recruitment and preoperative dilatation. | 14 days
Women with cervical dilatation ≥ 5 mm. | 14 days
Acceptability. | 14 days
Number of dilatations judged as "difficult." | 14 days
Frequency of complications. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Britt-Ingjerd Nesheim, MD, PhD, Study Chair — University of Oslo
Locations (1):
- Gynaecological Department, Ullevål University Hospital, Oslo, Norway